CLINICAL TRIAL: NCT01322009
Title: Overcoming Membrane Transporters to Improve CNS Drug Delivery
Brief Title: Overcoming Membrane Transporters to Improve CNS Drug Delivery - Improving Brain Antioxidants After Traumatic Brain Injury
Acronym: Pro-NAC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Robert Clark, MD, Critical Care Medicine, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NS069247; 1R01NS069247-01 (NIH)
Record Dates: First submitted 2011-03-22; First posted 2011-03-24 (Estimated); Results first posted 2016-08-15 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-07

CONDITIONS: Pediatric Traumatic Brain Injury
Keywords: Children; Brain injury; Trauma
MeSH Terms: conditions — Brain Injuries; Wounds and Injuries | interventions — Probenecid; Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug (Experimental): Probenecid and N-acetyl cysteine will be administered at standard doses for the first 4 days after TBI.
  Interventions: Drug: Probenecid and N-acetyl cysteine
- Placebo (Placebo Comparator): Placebos will be prepared for the two experimental drugs and administered at identical time periods.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Probenecid and N-acetyl cysteine — After obtaining written parental consent, patients will be randomized by the use of a blind envelope system to one of the following: to receive probenecid (initial: 25 mg/kg/dose; maintenance: 10mg/kg/dose 4 x per day for 11 doses) and NAC (initial: 140mg/kg/dose; maintenance: 70mg/kg/dose 6 x per day for 17 doses) or the placebo via nasogastric (NG) or orogastric (OG) tube for 3 days or to receive placebos.
  Arms: Drug
Drug: Placebo — After obtaining written parental consent, patients will be randomized by the use of a blind envelope system to one of the following: to receive probenecid (initial: 25 mg/kg/dose; maintenance: 10mg/kg/dose 4 x per day for 11 doses) and NAC (initial: 140mg/kg/dose; maintenance: 70mg/kg/dose 6 x per day for 17 doses) or the placebo via nasogastric (NG) or orogastric (OG) tube for 3 days. Placebo contents include equal volumes and dosing regimens of lactose powder (for opacity) suspended in Ora-Plus and normal saline.
  Other Names: Ora Plus
  Arms: Placebo

SUMMARY:
The overall purpose of this research study is to investigate the safety of pharmacological therapies that may potentially improve pediatric outcomes after traumatic brain injury. Traumatic brain injuries are the leading cause of death and disability among children and young adults.

Hypothesis: Combinational therapy with a membrane transporter and antioxidant are safe after TBI and can overcome barriers to the brain and synergistically improve bioavailability and efficacy the antioxidant content of the body and CNS after TBI.

DETAILED DESCRIPTION:
Specific Aim: Define the capacity of the combination of probenecid and NAC to safely and synergistically preserve levels of GSH and reduce oxidative stress in children with severe TBI. We will enroll 20 children age 2 to less than 18 years old (less than 216 months) after severe TBI in a randomized, controlled study of administration of the combinational therapy and test if the administration of these drugs is safe and if antioxidant reserve can be preserved within the serum and CSF.

Probenecid (at the same dose that is used as an adjunct to antibiotic therapy) and NAC (at the same dose that is used for acetaminophen-induced liver disease), or vehicles will be given for 3 days. The primary outcomes of the study will be the safety of drug administration and the CSF and serum levels anti-oxidant reserve (AOR), with the presumption that maintaining anti-oxidant levels within the brain may prove neuroprotective. Other secondary outcomes (CSF and serum probenecid, NAC, GSH and phenytoin concentrations) will also be tested. Adverse events occuring during treatment with these drugs after TBI will be monitored by a local Data Safety Monitoring Board.

ELIGIBILITY:
Inclusion Criteria:

* Children (age 2 - 18 y) with severe TBI (GCS < or = 8) with an externalized ventricular drain placed for measurement of intracranial pressure

Exclusion Criteria:

1. Brain dead on admission to ICU
2. Pregnancy
3. Contraindications to enteral medications
4. Contraindications to probenecid:

   * status epilepticus
   * blood dyscrasias
   * under 2 years-of-age
   * coadministration of salicylates
   * renal dysfunction or urate kidney stones
   * hypersensitivity to probenecid
5. Contraindications to N-acetylcysteine: hypersensitivity to N-acetylcysteine
6. Family unwilling to consent

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2011-03; Primary Completion 2013-12 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Bell, MD, Principal Investigator — University of Pittsburgh; Robert SB Clark, MD, Study Director — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Clark RSB, Empey PE, Kochanek PM, Bell MJ. N-Acetylcysteine and Probenecid Adjuvant Therapy for Traumatic Brain Injury. Neurotherapeutics. 2023 Oct;20(6):1529-1537. doi: 10.1007/s13311-023-01422-z. Epub 2023 Aug 18. PMID 37596428
- [Derived] Hagos FT, Empey PE, Wang P, Ma X, Poloyac SM, Bayir H, Kochanek PM, Bell MJ, Clark RSB. Exploratory Application of Neuropharmacometabolomics in Severe Childhood Traumatic Brain Injury. Crit Care Med. 2018 Sep;46(9):1471-1479. doi: 10.1097/CCM.0000000000003203. PMID 29742587
- [Derived] Clark RSB, Empey PE, Bayir H, Rosario BL, Poloyac SM, Kochanek PM, Nolin TD, Au AK, Horvat CM, Wisniewski SR, Bell MJ. Phase I randomized clinical trial of N-acetylcysteine in combination with an adjuvant probenecid for treatment of severe traumatic brain injury in children. PLoS One. 2017 Jul 7;12(7):e0180280. doi: 10.1371/journal.pone.0180280. eCollection 2017. PMID 28686657

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children 2-18 years-of-age after severe TBI (Glasgow Coma Scale [GCS] score ≤8) recruited from November 2011-September 2013 at a single, tertiary Children's Hospital.
Period: Overall Study
Arm/Group | Drug | Placebo
Started | 7 | 7
Completed | 7 | 4
Not Completed | 0 | 3
Not completed — Death | 0 | 1
Not completed — Adverse Event | 0 | 1
Not completed — ng tube discontinued | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Drug | Placebo | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 7 | 14
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.6 (4.9) | 9.7 (5.7) | 9.1 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 6 | 4 | 10
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Adverse Events
Description: The number of patients experiencing one or more of the following adverse events:
  Acute renal failure Anaphylaxis Acute respiratory distress syndrome Intracranial infection/abscess Arrhythmia, atrial Arrhythmia, ventricular Bradycardia Cardiac arrest Catheter positive culture Cerebrospinal fluid leak Decubitis Deep vein thrombosis Diabetes Insipidus Emesis Extraaxial hematoma Gastrointestinal bleed Gastritis Hematuria Hemorrhage, other Hemoperitonium Hemothorax Hepatitis Hydrocephalus Hypotension Hypoxemia Infection, other Intraparenchymal hemorrhage Intraventricular hemorrhage Meningitis/ventriculitis Multiorgan dysfunction syndrome Myocardial ischemia Pancreatitis Pericarditis Peritonitis Pneumothorax Pulmonary edema Pulmonary embolism Respiratory arrest Seizures Sepsis Syndrome of inappropriate antidiuretic hormone Transtentorial herniation Withdrawal of Life Support Other SAE causing re-hospitalization Other SAE
Time Frame: 14 days after drug administration
Measure: Number; unit: participants
Arm/Group | Drug | Placebo
Number analyzed (Participants) | 7 | 7
participants | 0 | 2

2. Secondary Outcome: Antioxidant Reserve
Description: Antioxidant reserves in CSF and serum will be calculated in both treatment arms and compared.
Time Frame: Within 5 days of injury
Measure: Mean (Standard Error); unit: reactive oxygen species scavenged
Arm/Group | Drug | Placebo
Number analyzed (Participants) | 7 | 7
reactive oxygen species scavenged | 751 (85) | 735 (117)
Statistical Analysis 1: Comparison: Drug vs Placebo; Test type: Superiority or Other; p > 0.05, ANOVA; Analysis run over study period but data entered only for the 6 h time point

ADVERSE EVENTS:
Arm/Group | Drug | Placebo
Serious Adverse Events (participants affected / at risk) | 0/7 | 1/7
Other Adverse Events (participants affected / at risk) | 0/7 | 1/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug (N=7) | Placebo (N=7)
death (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug (N=7) | Placebo (N=7)
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes